CLINICAL TRIAL: NCT04642768
Title: Treatment With the Ketone Body 3-hydroxybutyrate in Patients With Cardiogenic Shock
Acronym: KETO-SHOCK1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristoffer Berg-Hansen, Principal Investigator, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KETO-SHOCK 1-10-72-209-20
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Cardiogenic Shock
Keywords: Ketone bodies; β-hydroxybutyrate
MeSH Terms: conditions — Shock, Cardiogenic | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-Hydroxybutyrate treatment (Experimental): KetoneAid Ketone Ester 0,5g/kg (max. 50g) bolus
  Interventions: Dietary Supplement: KetoneAid Ketone Ester
- Placebo Treatment (Placebo Comparator): Maltodextrin-base isocaloric placebo
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: KetoneAid Ketone Ester — Commercially available ketone supplement
  Arms: 3-Hydroxybutyrate treatment
Dietary Supplement: Maltodextrin — Commercially available maltodextrin supplement
  Arms: Placebo Treatment

SUMMARY:
Background Cardiogenic shock is a life-threatening state of acute heart failure with severely depressed blood pressure and organ perfusion. The 30-day mortality is reported as high as 50%. To date, no randomized trial has documented a survival benefit of any medical treatment in this patient group. In a first-in-man study the investigators have recently discovered that treatment with ketone bodies increases cardiac output by 2 liters per minute.

Objective The present study aims to examine the direct effects of ketone body supplements on the heart function in patients hospitalized with cardiogenic shock. Also, the aim is to determine the relative need for medical circulatory support following ketone body supplement.

Design A randomized double-blind cross-over study of the hemodynamic effect of enteral ketone ester versus placebo in 12 patients with cardiogenic shock

Methods Right heart catheterization will be installed to monitor cardiac pressures and output. The investigators will observe heart function with transthoracic echocardiography. Blood- and urine samples will be analyzed for electrolytes, energy substrates and vasoactive substances. Organ perfusion is to be examined by renal ultrasonography and near-infrared spectroscopy for measuring cerebral and peripheral circulation.

Perspectives This investigation may grant essential knowledge on ketosis in cardiogenic shock. This may lead to larger clinical trials, and hopefully a new and better treatment for patients with cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing treatment with inotropes and/or vasopressors because of cardiogenic shock as judged by the clinicians
* Patients are required at some point in time to have had > 1 of the following: systolic blood pressure < 90 mmHg; arterial blood lactate ≥ 2.5mmol/l; organ hypoperfusion (e.g. urinary output < 0.5 ml/kg/hour or SvO2 <55% with normal PaO2 and Hgb)
* LVEF < 40%
* Age ≥ 18 years

Exclusion Criteria:

* Other primary causes of shock (hypovolemia, hemorrhage, severe infection or sepsis, pulmonary embolism or anaphylaxis),
* Shock due to mechanical complication to myocardial infarction (papillary muscle rupture, rupture of the ventricular septum or rupture of free wall)
* INTERMACS level 1 or 2 [18] with unstable or sliding hemodynamics on inotropes/vasopressors
* Use of or probable need for mechanic circulatory support (e.g. left ventricular assistant device, IMPELLA, extracorporeal membrane oxygenation)
* Recent post-cardiotomy cardiogenic shock (defined as thoracic surgery with the last 3 days)
* Inability to position a nasogastric tube
* Severe gastroparesis or abdominal distension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Cardiac Output (L/min) area under curve | 3 hours
  Right Heart Catheterization (by thermodilution)

SECONDARY OUTCOMES:
Cardiac output (L/min) | 1 hour
  Right Heart Catheterization (by thermodilution)
Left Ventricular Filling Pressure (mmHg) area under curve | 3 hours
  Right Heart Catheterization
Cardiac Power Output (W) area under curve | 3 hours
  mean arterial pressure x cardiac output/451
Mixed Venous Saturation (%) area under curve | 3 hours
  Right Heart Catheterization
Left Ventricular Ejection Fraction (%) area under curve | 3 hours
  Echocardiography
Hourly urinary output (mL/hour) area under curve | 3 hours
Renal Perfusion (mL/min) | 1 hours
  Renal doppler ultrasound
Arterial Lactate (mmol/L) area under curve | 3 hours
  Arterial blood gas measurements
Cumulative doses of inotropes and vasopressors during the 3 hour studyperiod | 3 hours
Cerebral Perfusion area under curve | 3 hours
  Near-infrared spectroscopy
Peripheral Perfusion area under curve | 3 hours
  Near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berg-Hansen K, Christensen KH, Gopalasingam N, Nielsen R, Eiskjaer H, Moller N, Birkelund T, Christensen S, Wiggers H. Beneficial Effects of Ketone Ester in Patients With Cardiogenic Shock: A Randomized, Controlled, Double-Blind Trial. JACC Heart Fail. 2023 Oct;11(10):1337-1347. doi: 10.1016/j.jchf.2023.05.029. Epub 2023 Jul 12. PMID 37452805